CLINICAL TRIAL: NCT06800495
Title: Development of THALEA (Thalassemia Education and Awareness) Kit and a Cluster Randomised Control Trial to Evaluate Its Effectiveness on Knowledge, Attitude, and Intention Regarding Premarital Thalassemia Screening Among Private Secondary School Students of Klang Valley, Malaysia
Brief Title: Development of THALEA Kit and Its Impact on Knowledge, Attitude, and Intention for Premarital Thalassemia Screening
Acronym: THALEA
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Teknologi Mara (Other)
Responsible Party: Principal Investigator, Maisarah binti Noor Anwar, DR, Universiti Teknologi Mara
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: THALEA; Other funds (Other: UiTM)
Record Dates: First submitted 2025-01-16; First posted 2025-01-30 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: Thalassemia
Keywords: Thalassemia; Educational intervention; secondary school students; THALEA; Thalassemia awareness; Premarital Thalassemia screening; Thalassemia education; thalassemia educational intervention; high school students; Malaysia; knowledge, attitude and intention
MeSH Terms: conditions — Thalassemia; Behavior | interventions — Receptor Protein-Tyrosine Kinases

STUDY DESIGN:
Intervention Model Description: THALEA (Thalassemia education and awareness) Kit is an educational intervention for secondary school students that is developed according to the theory of planned behaviour. It is to be delivered to high school students by a medical practitioner
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention arm (Experimental): vii. The intervention group will receive THALEA along with a basic family health education. THALEA's session comprises a face-to-face verbal presentation facilitated by the primary researcher, featuring an engaging interactive seminar and on-screen games. Following this, participants will be presented with 3-5-minute videos and pictorial materials, fostering two-way discussions. Subsequently, a softcopy of the THALEA kit will be distributed to the teacher in charge via email or WhatsApp after the seminar for further dissemination. The students will receive THALEA's brochures.
  Interventions: Behavioral: THALEA (Thalassemia Education and Awareness) Kit
- Comparison arm (Active Comparator): viii. The comparison group will only receive a basic family health education in which it is the usual family health education given by the MOH, usually delivered by a medical officer, to fourth form students at government schools prior to the thalassemia screening programme. It will consist of a delivery of a PowerPoint presentation and videos, that will be obtained from government public health clinics in Klang Valley.
  Interventions: Behavioral: Basic thalassemia and family health education

INTERVENTIONS:
Behavioral: THALEA (Thalassemia Education and Awareness) Kit — By using the opinions obtained by the experts, THALEA's content will then be designed using the Theory of Planned Behaviour (TPB) by Ajzen and Fishbein.
  Development of THALEA:
  • Language: Malay and English.
  • Contents of the THALEA kit: i. PowerPoint or Canva presentations with discussion prompts (softcopy form) ii. Links/joining codes to free educational game platforms such as Kahoot or Quizziz iii. Videos - convey messages on thalassemia awareness and screening importance.
  iv. Illustrated guides/brochures - to provide step-by-step tutorials on how to get thalassemia screening in both the public and private healthcare.
  • Developer would be the main researcher with aid from: i. Illustrator ii. Video graphic designer iii. Influencers
  • Delivery of THALEA to students by: i. Medical personnel
  Other Names: THALEA
  Arms: Intervention arm
Behavioral: Basic thalassemia and family health education — They are basic family health education in which it is the usual family health education given by the MOH, usually delivered by a medical officer, to fourth form students at government schools prior to the thalassemia screening programme. It will consist of a delivery of a PowerPoint presentation and videos, that will be obtained from government public health clinics in Klang Valley.
  Arms: Comparison arm

SUMMARY:
Thalassemia, a common genetic disease, is often overlooked compared to infectious diseases like HIV, despite its significant effects for families planning to have children. Thalassemia carriers are frequently asymptomatic, but when two carriers marry, there is a 25% chance of having a child with a severe form of the disease. Although screening programs exist, the number of symptomatic thalassemia major continues to increase, and current treatments are primarily symptomatic, merely prolonging survival rather than curing it.

In Malaysia, while HIV testing before marriage is mandatory, thalassemia screening is not. Presently, thalassemia screening and awareness programs are offered to fourth-form students in government schools only. Hence, there is a need to complement existing national screening efforts by creating a standardized thalassemia awareness program that can be effectively implemented across diverse educational institutions.

Our main objective is to develop and validate the THALEA (Thalassemia education and awareness) kit and evaluate its effectiveness among secondary school students in Klang Valley, Malaysia. We hope that with this intervention, high school students are be able to increase their awareness and knowledge, instil a positive attitude and have that intention to do a pre-marital thalassemia screening at any healthcare facility in our country. This can facilitate early detection and timely counselling to reduce the risk of having children with severe thalassemia.

Delivery of the intervention:

i. Schools will be approached by letter, followed by a phone call and a visit. ii. Consent forms will be given for parents to sign. iii. All fourth form students at the school will be invited to participate in the study, excluding those who meet the exclusion criteria.

iv. THALEA will be delivered by a face-to-face method between the main researcher and the students.

v. Frequency of delivery - one time only vi. Duration of intervention - 2-3 hours. vii. The intervention group will receive THALEA along with a basic family health education. THALEA's session comprises a face-to-face verbal presentation facilitated by the primary researcher, featuring an engaging interactive seminar and on-screen games. Following this, participants will be presented with 3-5-minute videos and pictorial materials, fostering two-way discussions. Subsequently, a softcopy of the THALEA kit will be distributed to the teacher in charge via email or WhatsApp after the seminar for further dissemination. The students will receive THALEA's brochures.

viii. The comparison group will only receive a basic family health education in which it is the usual family health education given by the MOH, usually delivered by a medical officer, to fourth form students at government schools prior to the thalassemia screening programme. It will consist of a delivery of a PowerPoint presentation and videos, that will be obtained from government public health clinics in Klang Valley.

We will use a self-administered questionnaire designed and validated to assess knowledge, attitude, and intention regarding premarital thalassemia screening among youths at three different time points which are during pre-assessment (t0), immediate post-assessment (t1), and 2 weeks post assessment (t2)

ELIGIBILITY:
Inclusion Criteria:

* Malaysians.
* Fourth form students.
* Able to read and write in either Malay or the English language.

Exclusion Criteria:

* Those who have previously undergone thalassemia screening
* Identified as thalassemia carriers
* Without parental consent or assent
* Has first-degree relatives diagnosed with thalassemia

Ages: 15 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 148 (Actual)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Knowledge and attitude score | i. All students will be given 5 minutes to fill in their demographic information ii. Then 10 to 15 minutes will be given to answer the questionnaire at three different time points which are during pre-assessment (t0), immediate post-assessment (t1), and
  Knowledge and attitude score will be calculated by using the filled in self-administered questionnaire designed and validated to assess knowledge, attitude, and intention regarding premarital thalassemia screening among youths

SECONDARY OUTCOMES:
Intention regarding premarital thalassemia screening | i. All students will be given 5 minutes to fill in their demographic information ii. Then 10 to 15 minutes will be given to answer the questionnaire at three different time points which are during pre-assessment (t0), immediate post-assessment (t1), and
  This will also be calculated using the same questionnaire.

CONTACTS AND LOCATIONS:
Locations (1):
- University Teknologi MARA, Sungai Buloh, Selangor, Malaysia

IPD SHARING:
Plan to Share IPD: No